CLINICAL TRIAL: NCT03141957
Title: Hypermetabolism in the Elderly Lung Cancer Patient
Acronym: HELP
Status: Completed | Type: Observational
Sponsor: University of Paris 5 - Rene Descartes (Other)
Responsible Party: Principal Investigator, Guillaume Ulmann, Doctor, University of Paris 5 - Rene Descartes
Other Study IDs: LBN001
Record Dates: First submitted 2017-04-28; First posted 2017-05-05 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Non-small Cell Lung Carcinoma
Keywords: Aging; Hypermetabolism
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Young patients: Patients with non-small cell lung carcinoma younger than 75y
- Elderly patients: Patients with non-small cell lung carcinoma aged 75 or more

SUMMARY:
Aging and cancer are two conditions associated with extensive metabolic changes that can cause malnutrition. However, the clinical features and the underlying mechanisms leading to malnutrition are different in these two cases. We therefore wonder how age can influence the metabolic response to cancer.

DETAILED DESCRIPTION:
During aging, among other physiological modifications, inactivity and insulin resistance cause a progressive muscle loss associated with a decrease in resting energy expenditure (REE). In cancer, loud inflammation background also provokes a decrease in muscle mass as well as in fat mass. However, previous studies reported an increased REE, termed hypermetabolism, probably linked to inflammation.

Data concerning response to aggression in the elderly patient is scarce and even inexistent when it comes to cancer. The investigators hypothesize that the mitochondrial dysfunction that comes with aging and that decreases the ATP rendering per unit of energy-producing nutrient oxidized increases the amount of nutrient to be consumed in order to sustain to energy needs. Therefore, in this situation, elderly patients could have a higher rate or degree of hypermetabolism than younger patients.

The primary objective of this study is to assess the effect of aging on the metabolic response to cancer assessed by resting energy expenditure measured by indirect calorimetry corrected by whole body fat free mass calculated from single slice CT imaging at the third lumbar vertebra.

The secondary objective of this study is to point out some inflammatory or endocrine determinants of these energy metabolism changes in the cancer patient.

Non-small cell lung carcinoma seems to be a relevant choice for this study because it is frequently associated with cachexia and the literature reports a high rate of hypermetabolism in this cancer.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung carcinoma

Exclusion Criteria:

* Imbalanced Diabetes
* Imbalanced dysthyroidia
* Surgery within two month prior inclusion
* Any chronic auto-immune or inflammatory disease

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population is selected from the patients coming for their one-day pre-treatment evaluation at the oncology ward of the Cochin Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Measured resting energy expenditure (mREE) in kilocalorie per day | Day 0
  Energy expenditure is measured by indirect calorimetry.

SECONDARY OUTCOMES:
Blood C-Reactive Protein in milligram per milliliter | Day 0
  Inflammatory status
Blood Interleukine-6 in picogram per milliliter | Day 0
  Inflammatory status
Blood Tumor Necrosis Factor alpha in picogram per milliliter | Day 0
  Inflammatory status
Blood Insulin in milliunit per liter | Day 0
  Endocrine Status - Glucose Homeostasis
Blood ultra-sensitive Thyroid Stimulating Hormone in milliunit per liter | Day 0
  Endocrine Status - Thyroid Function
Blood Insulin-like Growth Factor 1 in nanogram per liter | Day 0
  Endocrine Status - Somatotropic axis
Blood Glucose in millimole per liter | Day 0
  Endocrine Status
Homeostasis Model assessment of Insulin resistance | Day 0
  Aggregates blood Insulin and glucose level as an insulin resistance score
Lean Body Mass in kilogram | Day 0
  Estimated from muscular area at the third lombular vertebra from CT-scan
energy intake in kilocalorie per day | Day 0
  Estimated by a qualified dietetican
Albumin in gram per liter | Day 0
  Nutritional Satus
Transthyretin in gram per liter | Day 0
  Nutritional Satus
Predicted resting energy expenditure (HB) in kilocalorie per day | Day 0
  REE estimated with Harris & Benedict Formula
Percentage of estimated energy expenditure | Day 0
  Percentage of HB : (mREE/HB) x 100

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Cochin, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulmann G, Jouinot A, Tlemsani C, Curis E, Kousignian I, Neveux N, Durand JP, Goldwasser F, Cynober L, De Bandt JP. Lean Body Mass and Endocrine Status But Not Age Are Determinants of Resting Energy Expenditure in Patients with Non-Small Cell Lung Cancer. Ann Nutr Metab. 2019;75(4):223-230. doi: 10.1159/000504874. Epub 2019 Dec 19. PMID 31865308